CLINICAL TRIAL: NCT06105424
Title: BRP1602: Evaluation of Technical and Logistical Feasibility to Measure Lung Permeability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BRP1602
Record Dates: First submitted 2022-08-04; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2022-08

CONDITIONS: Tobacco Use; Smoking; Smoking, Tobacco
MeSH Terms: conditions — Tobacco Use; Smoking; Tobacco Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Smokers (Experimental): Someone who exclusively smokes 10 - 20 combustible filtered cigarettes per day (CPD) 83 - 100 mm in length, non-menthol or menthol, for at least 3 years prior to Screening.
  Interventions: Procedure: Lung Permeability Assessment
- Moist Snuff Consumers (Experimental): Someone who exclusively consumes ≥ 1 can of moist snuff per week for at least 6 months prior to Screening.
  Interventions: Procedure: Lung Permeability Assessment
- Vapers (Experimental): Someone who exclusively uses a nicotine-containing "cig-a-like" and/or tank system daily for at least 3 months prior to Screening.
  Interventions: Procedure: Lung Permeability Assessment
- Non-Tobacco Consumers (Experimental): Someone who has used no tobacco or nicotine-containing products for at least the past 5 years prior to Screening and do not plan to use any tobacco or nicotine-containing products throughout the study.
  Interventions: Procedure: Lung Permeability Assessment

INTERVENTIONS:
Procedure: Lung Permeability Assessment — A gamma camera will be used to scintigraphically monitor the clearance of an inhaled radiolabeled tracer molecule from the lungs into the blood. Clearance will be monitored for 60 minutes. The rate of clearance of radioactivity will serve as an index of alveolar epithelial permeability.

SUMMARY:
This will be a single-center, single-blind, four-cohort, 22-day ambulatory study during which up to 24 healthy adult subjects [6 smokers (SMK), 6 moist snuff consumers (MSC), 6 vapers (VAP), and 6 non-tobacco consumers (NTC)] will complete 3 measurements of lung permeability. Nasal epithelial cells, sputum, and blood samples will also be collected for current and future biomarker research.

DETAILED DESCRIPTION:
Test Visit 1 will consist of sampling for nasal epithelial cells, sputum, and blood. Additional subjects ("alternates") may be required to complete these procedures to better ensure that 24 subjects are available to complete the lung permeability assessments. During Test Visits 2, 3, and 4, subjects will provide additional blood samples and will complete the lung permeability procedure. A solution containing approximately 40 mCi of a radiolabeled tracer molecule (99mTc-DTPA) will be loaded into a radioaerosol administration system and subjects will breathe the aerosol over approximately 3 minutes, depositing approximately 1 mCi into the lungs (effective dose of approximately 0.3 rem). Subjects will lie supine in front of a gamma counter and a series of images will be obtained over 60 minutes, from which the 99mTc-DTPA clearance rate from the lungs will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 30 and 50 years, inclusive.
2. Subjects met one (a, b, c, or d) of the following tobacco or non-tobacco use conditions based on self-report:

   1. SMK who exclusively smoked 10 - 20 combustible filtered cigarettes per day (CPD) 83 - 100 mm in length, non-menthol or menthol, for at least 3 years prior to Screening. Brief periods of abstinence more than 30 days prior to Screening due to illness, quit attempt, or clinical study participation were allowed at the discretion of the Investigator.
   2. MSC who exclusively consumed ≥ 1 can of moist snuff per week for at least 6 months prior to Screening. Brief periods of abstinence more than 30 days prior to Screening due to illness, quit attempt, or clinical study participation were allowed at the discretion of the Investigator.
   3. VAP who exclusively used a nicotine-containing "cig-a-like" and/or tank system daily for at least 3 months prior to Screening. Subjects reported using only products with the characterizing flavors of tobacco, menthol, or fruit (e.g., berry, strawberry, blueberry, banana). Brief periods of abstinence more than 30 days prior to Screening due to illness, quit attempt, or clinical study participation were allowed at the discretion of the Investigator.
   4. NTC who had used no tobacco or nicotine-containing products for at least the past 5 years prior to Screening and did not plan to use any tobacco or nicotine containing products throughout the study.
3. Subjects met one (a, b, c, or d) of the following conditions:

   1. SMK had an ECO ≥ 15 ppm and ≤ 100 ppm and had a positive urine cotinine test (> 500 ng/mL).
   2. MSC had an ECO ≤ 5 ppm and had a positive urine cotinine test (> 500 ng/mL).
   3. VAP had an ECO ≤ 5 ppm and had a positive urine cotinine test (> 500 ng/mL).
   4. NTC had an ECO ≤ 5 ppm and had a negative urine cotinine test (≤ 200 ng/mL).
4. Generally healthy (i.e., free of any acute or chronic health conditions in the opinion of the Investigator).
5. Females had a negative serum pregnancy test result.
6. Subjects were able to read, understand, and willing to sign an ICF and complete questionnaires written in English.
7. Subjects were able to safely perform the required study procedures, as determined by the Investigator.
8. Females of childbearing potential were willing to use a form of contraception acceptable to the Investigator for the timing as noted below through study discharge. Examples of acceptable forms of contraception included, but were not limited to, the following.

   1. Surgeries:

      * Hysterectomy at least 6 months prior to Test Visit 1.
      * Bilateral oophorectomy at least 6 months prior to Test Visit 1.
      * Bilateral tubal ligation at least 6 months prior to Test Visit 1.
   2. Transcervical sterilization at least 6 months prior to Test Visit 1.
   3. Hormonal birth control at least 3 months prior to Test Visit 1.
   4. Non-hormonal intrauterine device (IUD) at least 3 months prior to Test Visit 1.
   5. Double barrier methods (e.g., condom and spermicide) at least 14 days prior to Test Visit 1.
   6. Abstinence at least 14 days prior to Test Visit 1.
   7. Vasectomized partner was acceptable birth control for females provided the surgery was performed at least 6 months prior to Test Visit 1.
   8. Postmenopausal at least 1 year prior to Test Visit 1 and confirmed by FSH > 40 mIU/mL.
   9. Non-vasectomized male subjects agreed to use a highly effective method of birth control (e.g., double-barrier method) with partners of childbearing potential and to not donate sperm during the study and for 90 days after the final administration of 99mTc-DTPA.

Exclusion Criteria:

1. Subjects who met one of the following based upon their cohort:

   1. For SMK, use of any tobacco- or nicotine-containing products (e.g., e-cigs, moist snuff, chewing tobacco, nicotine replacement therapy (NRT), tobacco cigarettes that are heated but not burned, dissolvable nicotine products) other than combustible cigarettes within 30 days prior to Screening. NOTE: Subjects who smoked ≤ 6 cigars in the past 12 months prior to Screening were NOT excluded. Subjects who received short-term administration of or used a NRT as a temporary bridging treatment/aid were NOT excluded.
   2. For MSC, use of any tobacco- or nicotine-containing products (e.g., combustible or heated cigarettes, e-cigs, chewing tobacco, NRTs, dissolvable nicotine products) other than moist snuff within 30 days prior to Screening or regular exposure to cigarette smoke within 60 days prior to Screening (e.g., lived with a smoker who smoked in the home). NOTE: Subjects who received short-term administration of or used a NRT as a temporary bridging treatment/aid were NOT excluded.
   3. For VAP, use of any tobacco- or nicotine-containing products (e.g., combustible or heated cigarettes, moist snuff, chewing tobacco, NRTs, dissolvable nicotine products) other than nicotine-containing vaping products within 30 days prior to Screening or regular exposure to cigarette smoke within 60 days prior to Screening (e.g., lived with a smoker who smoked in the home). NOTE: Subjects who received short-term administration of or used a NRT as a temporary bridging treatment/aid were NOT excluded.
   4. For NTC, use of any tobacco- or nicotine-containing products (e.g., combustible or heated cigarettes, e-cigs, moist snuff, chewing tobacco, NRTs, dissolvable nicotine products) within 5 years prior to Screening or regular exposure to cigarette smoke within 60 days prior to Screening (e.g., lived with a smoker who smoked in the home).
2. Clinically significant or unstable/uncontrolled acute or chronic medical conditions, as determined by the Investigator, that precluded a subject from participating safely in the study (e.g., uncontrolled hypertension, asthma or other lung disease, or cardiac disease) based on safety assessments such as clinical laboratory tests, medical history, and physical/nasopharyngeal examinations.
3. History, presence, or clinical laboratory test results indicating diabetes.
4. Presence of environmental allergies that result in allergic rhinitis which had been treated with any medication within 2 weeks of sample collection.
5. Observed or report of a heavy cough that precluded a subject from successfully completing the lung permeability assessment.
6. Use of any NRT or smoking cessation medication (e.g., nicotine gum, lozenge, or patch; varenicline [Chantix®], bupropion [Wellbutrin®, Zyban®]) within 30 days prior to Screening through completion of the study.
7. A female who was pregnant, planned to become pregnant during the course of the study, or was breast feeding.
8. Females ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
9. Post-bronchodilator FEV1:FVC ratio < 0.7 and FEV1 < 80% of predicted.
10. Post-bronchodilator FEV1:FVC ratio < 0.75 and FEV1 increase ≥ 12% (or > 200 mL) from pre- to post-bronchodilator.
11. Systolic blood pressure > 150 mmHg or diastolic blood pressure > 95 mmHg.
12. Fever (i.e., body temperature > 100.5°F).
13. Body mass index (BMI) < 18.5 or > 40.0 kg/m2.
14. Estimated creatinine clearance (by Cockcroft-Gault equation) < 80 mL/minute.
15. Positive urine drug screen or alcohol test.
16. Unwilling to follow study guidelines.
17. Known history of any condition that may cause nose bleeds.
18. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
19. Postponing a decision to quit tobacco product use (defined as planning a quit attempt within 30 days of Screening) to participate in this study or previous attempt within 30 days prior to Screening.
20. Participation in another clinical trial within 30 days prior to the first Test Visit. The 30 day window for each subject was derived from the date of the last study event in the previous study to the first Test Visit of the current study.
21. Participation in another clinical trial in which a radiolabeled compound was administered within 1 year prior to the first Test Visit.
22. Had received radiolabeled substances or had been exposed to radiation sources over the past 12 months or was likely to receive radiation exposure or radioisotopes within the next 12 months, such that participation in this study would increase the subject's total exposure beyond the recommended levels considered safe (i.e., weighted annual limit recommended by the International Commission on Radiological Protection of 3000 mrem).

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09-24 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Lung Permeability Feasibility | 60 minutes
  Assess the technical and logistical feasibility of conducting a clinical evaluation of lung permeability as a potential biomarker of effect of tobacco use.The outcome measure of this method development study: "the half-life (T 1/2) of inhaled 99mtechnetium diethylenetriaminepentaacetic acid (99mTC-DTPA) in lungs of study subjects by scintigraphy."

CONTACTS AND LOCATIONS:
Overall Officials: Patrudu Makena, PhD, Study Director — RAIS
Locations (1):
- Celerion, Inc., Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No